CLINICAL TRIAL: NCT02609529
Title: Double-Blind, Randomized Pilot Study Evaluating Oral Serum-Derived Bovine Immunoglobulin Protein Isolate (SBI) on Nutritional Status in Children With Diarrhea-Predominant Irritable Bowel Syndrome (d-IBS)
Brief Title: SBI in Children With d-IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: Entera Health, Inc (Industry)
Responsible Party: Principal Investigator, Rachel Herdes, Co-investigator, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB 8847
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Pediatrics; Nutrition
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SBI (Experimental): Entergam 10 g/day PO
  Interventions: Other: Medical Food
- Placebo (Placebo Comparator): Placebo 10 g/day PO
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Medical Food — Serum-derived bovine immunoglobulin protein isolate will be supplied by EnteraHealth. The product is manufactured in accordance with Good Manufacturing Practice (GMP) and U.S. Food and Drug Administration (FDA) guidelines for medical food ingredients (21 CFR Part 110). Serum-derived bovine immunoglobulin protein isolate (SBI) is generally recognized as safe (GRAS). The FDA has reviewed the safety dossier for SBI as a medical food product.
  Other Names: Enteragam
  Arms: SBI
Other: Placebo
  Arms: Placebo

SUMMARY:
IBS is the most common diagnosis in new patients in our pediatric gastroenterology clinic, accounting for 36 % of all new patients. Pediatric IBS patients always have a problem with defecation, characterized either as diarrhea predominant or constipation predominant. About one third of pediatric IBS subjects have d-IBS. There are no FDA approved treatments for children with d-IBS. There is evidence that diarrhea predominant irritable bowel syndrome d-IBS may be caused by a mild inflammation in the intestinal lining. Oral serum-derived bovine immunoglobulin protein isolate (SBI) is a medical food, believed to treat mild inflammation in the small intestine associated with some cases of d-IBS, especially those arising after acute gastroenteritis. It improved pain and diarrhea in adults with d-IBS. Our aim is to determine if SBI improves the number of spontaneous bowel movements in children with d-IBS.

DETAILED DESCRIPTION:
The objectives of the study are to determine whether there is improvement in gastrointestinal symptoms (i.e., number of spontaneous bowel movements. abdominal pain, stool consistency, reduction in stool number, flatulence, urgency, incontinence), in laboratory parameters, and/or in psychosocial measures in subjects with d-IBS receiving 3 weeks of SBI.

This is a randomized, double-blind, placebo-controlled, weighted, pilot study evaluating effects of SBI (10 g per day), in children or adolescents with d-IBS.

The primary outcome will be change in the number of spontaneous bowel movements from the screening week compared to the final week. This information is gathered as part of the daily diary questions.

Secondary clinical outcome variables will include changes in abdominal pain, stool consistency, flatulence, urgency, and incontinence. Further clinical outcome variables will be change in number of spontaneous bowel movements during each treatment week compared to the screening week. Stool consistency will be assessed with the Bristol Stool Form Scale. Secondary laboratory outcome variables will include changes in stool calprotectin, stool lactoferrin, erythrocyte sedimentation rate, C-reactive protein, and platelet count from the screening week and final week. Secondary psychosocial outcomes will include data from Pediatric Quality of Life Inventory for Gastrointestinal Symptoms, and the Pediatric Functional Disability Index.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females between 8 years and 18 years at the time of consent.
2. Able to obtain parental or legal guardian informed consent from subjects as applicable.
3. d-IBS determined by ROME III criteria. A Rome III diagnosis consists of recurrent abdominal pain or discomfort at least 2days/week in the last 3 months prior to enrollment associated with two or more of the following10:

1. Improvement with defecation 2. Onset associated with a change in frequency of stool 3. Onset associated with a change in form (appearance) of stool.

Exclusion Criteria:

1. Children taking pharmacologic treatment for d-IBS will be excluded.
2. Children who are unable to articulate symptoms of IBS will be excluded.
3. Non-English speaking children will be excluded.
4. Children with known allergy or hypersensitivity to beef or any component of SBI.
5. Pregnancy.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
Number of spontaneous bowel movements | 3 weeks
  The primary outcome will be change in the number of spontaneous bowel movements from the screening week compared to the final week. This information is gathered as part of the daily diary questions.

SECONDARY OUTCOMES:
Stool consistency | 3 weeks
  Bristol Stool Scale
Laboratory values | 3 weeks
  Stool calprotectin, stool lactoferrin, ESR, CRP, platelet count
Psychosocial | 3 weeks
  Pediatric Quality of Life Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hyman, MD, Principal Investigator — LSUHSC
Locations (1):
- Childrens Hospital, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Giannetti E, de'Angelis G, Turco R, Campanozzi A, Pensabene L, Salvatore S, de Seta F, Staiano A. Subtypes of irritable bowel syndrome in children: prevalence at diagnosis and at follow-up. J Pediatr. 2014 May;164(5):1099-1103.e1. doi: 10.1016/j.jpeds.2013.12.043. Epub 2014 Jan 31. PMID 24485818
- [Background] Camilleri M, Lasch K, Zhou W. Irritable bowel syndrome: methods, mechanisms, and pathophysiology. The confluence of increased permeability, inflammation, and pain in irritable bowel syndrome. Am J Physiol Gastrointest Liver Physiol. 2012 Oct;303(7):G775-85. doi: 10.1152/ajpgi.00155.2012. Epub 2012 Jul 26. PMID 22837345
- [Background] Asmuth DM, Ma ZM, Albanese A, Sandler NG, Devaraj S, Knight TH, Flynn NM, Yotter T, Garcia JC, Tsuchida E, Wu TT, Douek DC, Miller CJ. Oral serum-derived bovine immunoglobulin improves duodenal immune reconstitution and absorption function in patients with HIV enteropathy. AIDS. 2013 Sep 10;27(14):2207-17. doi: 10.1097/QAD.0b013e328362e54c. PMID 23660579
- [Background] Jiang R, Chang X, Stoll B, Fan MZ, Arthington J, Weaver E, Campbell J, Burrin DG. Dietary plasma protein reduces small intestinal growth and lamina propria cell density in early weaned pigs. J Nutr. 2000 Jan;130(1):21-6. doi: 10.1093/jn/130.1.21. PMID 10613760
- [Background] Bosi P, Casini L, Finamore A, Cremokolini C, Merialdi G, Trevisi P, Nobili F, Mengheri E. Spray-dried plasma improves growth performance and reduces inflammatory status of weaned pigs challenged with enterotoxigenic Escherichia coli K88. J Anim Sci. 2004 Jun;82(6):1764-72. doi: 10.2527/2004.8261764x. PMID 15217004
- [Background] Wilson D, Evans M, Weaver E, Shaw AL, Klein GL. Evaluation of serum-derived bovine immunoglobulin protein isolate in subjects with diarrhea-predominant irritable bowel syndrome. Clin Med Insights Gastroenterol. 2013 Dec 5;6:49-60. doi: 10.4137/CGast.S13200. eCollection 2013. PMID 24833942
- [Background] Walker LS, Greene JW. The functional disability inventory: measuring a neglected dimension of child health status. J Pediatr Psychol. 1991 Feb;16(1):39-58. doi: 10.1093/jpepsy/16.1.39. PMID 1826329
- [Background] Varni JW, Kay MT, Limbers CA, Franciosi JP, Pohl JF. PedsQL gastrointestinal symptoms module item development: qualitative methods. J Pediatr Gastroenterol Nutr. 2012 May;54(5):664-71. doi: 10.1097/MPG.0b013e31823c9b88. PMID 22008958